CLINICAL TRIAL: NCT04594499
Title: The Relationship Between Pericardial Fat Thickness and Arterial Stiffness in Heart Failure With Preserved Ejection Fraction Patients
Brief Title: The Relationship Between Pericardial Fat Thickness and Arterial Stiffness in HFpEF Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2020-10
Record Dates: First submitted 2020-10-15; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: epicardial fat tissue, arterial stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) was considered as a heterogeneous disease with multi-organ and multi-system design, which is related to various complications, such as hypertension, obesity and arteriosclerosis. Studies have found that hypertension and obesity are respectively associated with increased arterial stiffness. However, there is still no research investigating the the relationship between blood pressure and arterial stiffness in HFpEF patients with different levels of obesity.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) has typical symptoms and signs of heart failure with preserved ejection fraction (LVEF≥50%). Often associated with obesity, hyperlipidemia and other metabolic syndromes. At present, the incidence of HFpEF accounts for about 50% of heart failure, and it is increasing year by year. However, the specific pathogenesis of HFpEF is unknown, and there is a lack of effective diagnosis and treatment methods. A number of studies have shown that obesity is a unique pathophysiological phenotype of individuals with HFpEF, and the activation of inflammatory mediators is extremely prominent in the pathophysiological process of HFpEF. Therefore, we speculate that both obesity and inflammation are related to increased arterial stiffness.

Obesity is a heterogeneous disease. Certain ectopic fats, such as epicardial adipose tissue (EAT), may be related to obesity-related cardiovascular risks. EAT is a kind of visceral fat. Under pathological conditions, it releases factors harmful to the coronary artery and myocardium, and promotes the transition of EAT to a pro-inflammatory and pro-fibrotic phenotype. Brachial ankle pulse wave velocity (baPWV) is an indicator for evaluating arterial stiffness. It is a relatively simple, non-invasive method for detecting vascular compliance and an independent prediction of cardiovascular events in people without cardiovascular disease. Factors can be used to assess the risk of cardiovascular events. However, no relevant research has confirmed that pericardial fat can increase the arterial stiffness of HFpEF.

This study intends to observe the influence of pericardial fat on the arterial stiffness of HFpEF and explore the relationship between pericardial fat thickness and arterial stiffness of HFpEF, in order to assist the clinic in evaluating the vascular state of HFpEF patients faster and better, and to judge the prognosis. At the same time, EAT has the characteristics of fast metabolism, strong organ fat specificity, and simple measurement. It can also be used as a target for drug targeted therapy, opening up a new way for drug therapy of cardiometabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged >=18years old;
* Diagnosed with HFpEF.

Diagnostic criteria including:

1. left ventricular ejection fraction ≥50%；
2. with the symptoms and/or signs of heart failure；
3. BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL；
4. at least one additional criterion: relevant structural heart disease(LVH and/or LAE) or diastolic dysfunction

Exclusion Criteria:

* LVEF less than 45% at any time;
* Severe liver failure;
* Primary pulmonary hypertension;
* Age <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | On admission
  The arterial stiffness of HFpEF patients, for example brachial ankle pulse wave velocity, ardioankle vascular index and so on.
Epicardial Fat Tissue | On admission
  Epicardial Fat Tissue by cardiac color Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No